CLINICAL TRIAL: NCT01002313
Title: Effect of Prednisone on Peripheral Blood T-cell Function (Tregs and Th17) in Patients With Chronic Rhinosinusitis (CRS)
Brief Title: Effect of Prednisone onTregs and TH17
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 09-254-A
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-03

CONDITIONS: Chronic Rhinosinusitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- normal control
- Patient treatment group: Treatment with prednisone

SUMMARY:
The primary objective of this study is to see whether systemic corticosteroids (such as Prednisone) have an effect on the peripheral blood Treg and Th17 function in patients with CRS. Patients are taking prednisone as part of their routine medical care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CRS.
* A CT scan performed in the last year depicting the severity of the disease or nasal polyps on endoscopy.
* Symptomatic at the time of entry into the study as determined by scores ≥ 1.4 on the Rhinosinusitis disability index

Exclusion Criteria:

* Women who are pregnant or breastfeeding.
* Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study (heart, lung, kidney, diabetes, osteoporosis, cataracts, glaucoma, neurological, oncologic, liver disease or a contraindication to taking prednisone).
* Use of any other investigational agent in the last 30 days.
* Use of clinical drugs like antihistamines, leukotriene modifiers, intranasal steroids, systemic corticosteroids in the last 15 days or immunotherapy in the last year.
* Upper respiratory infection within 14 days of study start
* Smoking within the last 2 months.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with seasonal allergies taking prednisone and normal controls form the community.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-11; Primary Completion 2010-05 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Treg cell numbers | pre treatment vs post treatment

SECONDARY OUTCOMES:
Cytokine levels in cultured PBMCs | pre vs post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Naclerio, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Watanabe S, Pinto JM, Bashir ME, De Tineo M, Suzaki H, Baroody FM, Naclerio RM, Sharma S. Effect of prednisone on nasal symptoms and peripheral blood T-cell function in chronic rhinosinusitis. Int Forum Allergy Rhinol. 2014 Aug;4(8):609-16. doi: 10.1002/alr.21336. Epub 2014 Apr 21. PMID 24753507